CLINICAL TRIAL: NCT02600988
Title: Immunomodulatory Effect of Vitamin D in Allogenic Post-transplant
Acronym: Alovita-1
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Fundación Pública Andaluza para la gestión de la Investigación en Sevilla (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Alovita-1
Record Dates: First submitted 2015-06-09; First posted 2015-11-10 (Estimated); Last update posted 2015-11-10 (Estimated); Status verified 2015-11

CONDITIONS: Hematopoietic Stem Cell Transplantation
Keywords: Graft-Versus-Host-Disease; post-allogeneic transplant; haematopoietic progenitors
MeSH Terms: conditions — Graft vs Host Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Group 1: Control (No Intervention): Control group is composed by the first 50 patients included in the study. Those patients will not receive the treatment. Evaluations and follow-up will be the same as in the other groups.
- Group 2: 1000IU/day of Vitamine D (Experimental): It is composed by the following 50 patients joining the study. They will take 1000 IU of vitamin D once a day.
  Interventions: Drug: 1000IU/day of Vitamine D
- Group 3: 5000IU/day of Vitamine D (Experimental): It is composed by the last 50 patients joining the study. They will take 5000 IU of vitamin D once a day.
  Interventions: Drug: 5000IU/day of Vitamine D

INTERVENTIONS:
Drug: 1000IU/day of Vitamine D — Administration of a specified dose of Vitamine D
  Other Names: Vitamine D dose of 1000 international units (IU)
  Arms: Group 2: 1000IU/day of Vitamine D
Drug: 5000IU/day of Vitamine D — Administration of a specified dose of Vitamine D
  Other Names: Vitamine D dose of 5000 international units (IU)
  Arms: Group 3: 5000IU/day of Vitamine D

SUMMARY:
The purpose of this study is to determine whether vitamin D is effective in the prevention of graft-versus-host-disease after completion of allogeneic transplant.

DETAILED DESCRIPTION:
The allogeneic transplant of haematopoietic cell is the only treatment option for many malignant blood diseases. Unfortunately, the progression free survival and the quality of life of transplanted patients is limited due to the development of graft-versus-host-disease (GVHD).

The development of new prophylaxis strategies of GVHD based in the use of immunomodulator agents (allowing the generation of an immunotolerance state and avoiding the use of immunosuppression) is essential.

The GVHD is due to the cytotoxic effect of the donor lymphocytes T against healthy organs and tissues of the receptor. Calcineurin inhibitor combined with methotrexate or antibodies anti-lymphocytes T are used as standard prophylaxis. This type of antibodies has demonstrated efficacy to reduce GVHD, but have not increased survival due to increasing the risk of relapses and serious post-transplant infections.

Due to its interactions with VDR (vitamin D receptor) present in immune system cells, vitamin D is able to inhibit the activation of dendritic cells and the proliferation and production of cytokines by lymphocytes T. Based on this effect, the peri- and post- transplant administration of vitamin D might decrease the risk of GVHD in allogeneic transplanted patients, subsequently decreasing the immunosuppressant treatment requirements and improving the prognosis of those patients.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* The patient should accomplish all the criteria to proceed to an allogeneic transplant
* The patient or their legal guardians should signed the informed consent approved by the Ethics Committees of Clinical Trials

Exclusion Criteria:

* Hypercalcemia ≥ 10.5 mg/dl
* Renal insufficiency with creatinine level ≥ 2 x upper limit of normal (1,1 mg/dl)
* Participation in others Clinical Trials in which the intervention may affect the result of the study.
* Patients receiving GVHD immunoprophylaxis with thymoglobuline or GVHD prophylaxis including in vitro or in vivo lymphocytes T depletion (anti-lymphocyte T globulin, ALG)
* Patients receiving a transplant from an haploidentical donor

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2011-07; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Incidence/severity of Graft-Versus-Host-Disease | Day +150 post-transplant
  Number of cases of GVHD/Seriousness graded according to National Institutes of Health Consensus Development Project on Criteria for Clinical Trials in Chronic Graft-versus-Host Disease

SECONDARY OUTCOMES:
Serum levels of Th1/Th2 cytokines | Day -5 pre-transplant and +1, +7, +21,+56 and +100 post-transplant
  (IL-2, IL-4, IL-6, IL-10, tumor necrosis factor alfa (TNF)-α and interferon gamma (IFN-g)) are determined by flow cytometry using the BD Human Th1/Th2 Cytokine CBA
Dendritic cells | Day +21,+56 and +100 post-transplant
  The following markers were used to identify different subpopulations
  CD16-PB, CD45-V500, HLADR-FITC, BDCA-PE, CD11c-PerCP-Cy5.5, CD86-PE-Cy7, CD123-APC and CD14-APC-H7.
  Plasmacytoid dendritic cells: HLADR+ CD123++ CD11c- CD16- CD14- BDCA1- CD45+.
  Monocyte-derived dendritic cells: HLADR+ CD123+d CD11c+ CD16++ CD14-/+d BDCA- CD45+.
  Myeloid BDCA1 dendritic cells : HLADR+ CD123- CD11c+ CD16- CD14- BDCA+ CD45+
Subpopulations of lymphocytes | Day +21,+56 and +100 post-transplant
  To be identified using the combination CD19+CD8-FITC, CD3+CD56-PE, CD4- PerCP-Cy5.5, HLADR-APC T cells: CD3+ (CD3+CD4+CD8-, CD3+CD4-CD8+, CD3+CD4+CD8+, CD3+CD4-CD8+)
  B cells: CD19+ HLADR+
  NK cells: CD3- CD19- CD56+
  CD45RA-FITC and CCR7-PE were used to distinguish the repertory of naive/effector/memory of CD4 and CD8 cells.
  -naive T cells: CD45RA+CCR7+
  -effector T cells: CD45RA+CCR7-
  -central memory T cells: CD45RA-CCR7+
  -Peripheral memory T cells: CD45RA-CCR7-
Regulatory T cells | Day +21,+56 and +100 post-transplant
  after incubation of surface antigens (CD25-FITC, CD127-PE and CD4-PerCP-Cy5.5), cells were washed in PBS and then fixed and permeabilized with FoxP3 Staining Buffer Set (eBiosciences) for FOXP3 staining.
  phenotype of Treg: CD4+CD25+CD127-/+wFoxP3+
NK markers | Day +21,+56 and +100 post-transplant
  using the following combinations:
  CD94-FITC/CD56-PE/CD3-PerCP-Cy5.5/HLADR-APC
  CD11a-FITC/CD16-PE/CD3-PerCP-Cy5.5/CD56-APC
  CD158a-FITC/CD161-PE/CD3-PerCP-Cy5.5/CD56-APC
  CDNKB1-FITC/NKAT-PE/CD3-PerCP-Cy5.5/CD56-APC
  We identify NK cells with weak expression of CD56 (CD56 called " weak) and those expressing more intensely this marker CD56 "bright ". In addition the expression of different KIR receptor as CD158a , CD161 , and NKAT2 NKB1 were reported.
Activation of T cells | Day +21,+56 and +100 post-transplant
  Activation assays are performed on 500 µl of peripheral blood added in 48-well plates. Peripheral blood is stimulated or not with PMA (20µg/2ml) and ionomycin (0.91 µg/ml).
Peak Plasma Concentration (Cmax) of Vitamin D | Day -5 pre-transplant and +1, +7 and +21 post-transplant
  Peak Plasma Concentration (Cmax)
Area under the plasma concentration of Vitamin D | Day -5 pre-transplant and +1, +7 and +21 post-transplant
  Area under the plasma concentration versus time curve (AUC)
Bone densitometry changes carried out by protocol in post-transplant period | Day +150 post-transplant
  Treatment effect in the subsequent development of osteoporosis

CONTACTS AND LOCATIONS:
Overall Officials: José Antonio Pérez-Simón, MD-PhD, Study Chair — Head of haematology department
Locations (7):
- Spain (7):
  - Christelle Ferrà i Coll, Badalona, Barcelona
  - Carmen Martínez, Barcelona, Barcelona
  - David Valcárcel Ferreiras, Barcelona, Barcelona
  - Raquel Saldaña Moreno, Jerez de la Frontera, Cádiz
  - Manuel Jurado Chacón, Granada, Granada
  - Mª Ángeles Cuesta, Málaga, Málaga
  - Fermín Martín Sánchez- Guijo, Salamanca, Salamanca

REFERENCES:
- [Derived] Carrillo-Cruz E, Garcia-Lozano JR, Marquez-Malaver FJ, Sanchez-Guijo FM, Montero Cuadrado I, Ferra I Coll C, Valcarcel D, Lopez-Godino O, Cuesta M, Parody R, Lopez-Corral L, Alcoceba M, Caballero-Velazquez T, Rodriguez-Gil A, Bejarano-Garcia JA, Ramos TL, Perez-Simon JA. Vitamin D Modifies the Incidence of Graft-versus-Host Disease after Allogeneic Stem Cell Transplantation Depending on the Vitamin D Receptor (VDR) Polymorphisms. Clin Cancer Res. 2019 Aug 1;25(15):4616-4623. doi: 10.1158/1078-0432.CCR-18-3875. Epub 2019 May 1. PMID 31043390
- [Derived] Caballero-Velazquez T, Montero I, Sanchez-Guijo F, Parody R, Saldana R, Valcarcel D, Lopez-Godino O, Ferra I Coll C, Cuesta M, Carrillo-Vico A, Sanchez-Abarca LI, Lopez-Corral L, Marquez-Malaver FJ, Perez-Simon JA; GETH (Grupo Espanol de Trasplante Hematopoyetico). Immunomodulatory Effect of Vitamin D after Allogeneic Stem Cell Transplantation: Results of a Prospective Multicenter Clinical Trial. Clin Cancer Res. 2016 Dec 1;22(23):5673-5681. doi: 10.1158/1078-0432.CCR-16-0238. Epub 2016 Jun 29. PMID 27358490